CLINICAL TRIAL: NCT02489357
Title: A Pilot Study of MK-3475 With Cryotherapy for Men With Newly Diagnosed Oligo-metastatic Prostate Cancer
Brief Title: Pembrolizumab and Cryosurgery in Treating Patients With Newly Diagnosed, Oligo-metastatic Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1534; NCI-2015-00981 (Other: CTRP (Clinical Trial Reporting Program)); IRB00045444; MK-3475; P30CA006973 (NIH)
Record Dates: First submitted 2015-06-30; First posted 2015-07-03 (Estimated); Results first posted 2019-04-03 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cryosurgery; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pembrolizumab, cryosurgery) (Experimental): Patients receive standard of care degarelix SC once a month for 8 months. Within 1 month of receiving degarelix, patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Within 3 days of receiving pembrolizumab, patients undergo whole gland cryoablation of the prostate.
  Interventions: Procedure: Cryosurgery; Drug: Degarelix; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Procedure: Cryosurgery — Undergo whole gland cryoablation
  Other Names: CRYOABLATION; cryosurgical ablation
Drug: Degarelix — Given SC
  Other Names: FE200486; Firmagon
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This pilot phase II trial studies the side effects and how well pembrolizumab and cryosurgery work with short term androgen ablation to treat patients with prostate cancer that has traveled from the original tumor, through the body, and formed a small number of new tumors in other parts of the body (oligo-metastatic). Cryosurgery, also known as cryoablation or cryotherapy, kills tumor cells by freezing them. The process also incites an immune response within the ablated tumor. Giving monoclonal antibodies such as pembrolizumab which enhance a systemic anti-cancer immune response, may augment the effects of cryosurgery and increase tumor killing at distant (metastatic) sites.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess feasibility via the proportion of men reaching a low prostate-specific antigen (PSA) nadir (< 0.6 ng/ml) at 1 year.

II. Evaluate the safety of cryotherapy to the prostate combined with pembrolizumab.

TERTIARY OBJECTIVES:

I. To evaluate the effects of combination cryotherapy / pembrolizumab on programmed cell death 1 (PD-1) and programmed cell death 1 ligand 1 (PD-L1) expression in the prostate as assessed by biopsy performed 6 months post treatment.

OUTLINE:

Patients receive standard of care androgen ablation with degarelix subcutaneously (SC) once a month for 8 months. Within 1 month of receiving degarelix, patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Within 3 days of receiving the first dose of pembrolizumab, patients undergo whole gland cryoablation of the prostate.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically diagnosed oligo-metastatic prostate cancer; oligo-metastatic disease is defined to reflect men with low volume disease; specifically, oligo-metastatic disease is defined as less than 5 extra-pelvic metastases; metastatic lesions may be lymph nodes
* Be willing and able to provide written informed consent/assent for the trial
* Have available tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion
* Eastern Cooperative Oncology Group (ECOG) performance scale status of 0 or 1
* Demonstrate adequate organ function, all screening labs should be performed within 14 days of treatment initiation
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L
* Serum creatinine OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) =< 1.5 X upper limit of normal (ULN) OR >= 60 mL/min for subject with creatinine levels > 1.5 X institutional upper limit of normal (ULN)
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulant
* Have testosterone greater than 50 ng/dl
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has had a prior monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent; Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study; Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study; subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is expecting to father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-cluster of differentiation (CD)137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis c (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] (qualitative) is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment
* Has severe voiding symptoms (International Prognostic Scoring System [IPSS] > 20) or urinary retention requiring a catheter
* Has contraindications to cryotherapy of the prostate, including: previous transurethral prostatic resection (TURP) with persistent transurethral resection (TUR) defect, existing peri-anal or recto-urethral fistula, previous external beam radiation therapy or brachytherapy, coagulopathy, inability to tolerate anesthesia (spinal or general), inability to tolerate transrectal ultrasound (i.e. history of previous abdominal perineal resection)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Antonarakis, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ross AE, Hurley PJ, Tran PT, Rowe SP, Benzon B, Neal TO, Chapman C, Harb R, Milman Y, Trock BJ, Drake CG, Antonarakis ES. A pilot trial of pembrolizumab plus prostatic cryotherapy for men with newly diagnosed oligometastatic hormone-sensitive prostate cancer. Prostate Cancer Prostatic Dis. 2020 Mar;23(1):184-193. doi: 10.1038/s41391-019-0176-8. Epub 2019 Oct 14. PMID 31611635

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab, Cryosurgery)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab, Cryosurgery)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With PSA < 0.6 ng/mL
Time Frame: At 1 year
Population: Data was not collected in 1/12 participants due to lost to follow up before one year.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Cryosurgery)
Number analyzed (Participants) | 11
Participants | 5

2. Other Pre Specified Outcome: Expression of PD-1
Description: Number of participants with PD-1 expression in tumor tissue.
Time Frame: Baseline
Population: 1 participant refused biopsy. Only 2/11 samples were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Cryosurgery)
Number analyzed (Participants) | 2
Participants | 1

3. Other Pre Specified Outcome: Expression of PD-L1
Description: Number of participants with PD-L1 expression in tumor tissue.
Time Frame: Baseline
Population: 1 participant refused biopsy. Only 2/11 samples were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Cryosurgery)
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: up to 2 years
Arm/Group | Treatment (Pembrolizumab, Cryosurgery)
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Cryosurgery) (N=12)
Edema (Blood and lymphatic system disorders) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 3 (3)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Fatigue (General disorders) | 8 (8)
Hot flashes (Vascular disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 3 (3)
Injection site reaction (General disorders) | 3 (3)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Maculo-papular Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Mucositis (Gastrointestinal disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Penile pain (Reproductive system and breast disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Groin Pain (Gastrointestinal disorders) | 3 (3)
Night sweats (Metabolism and nutrition disorders) | 1 (1)
Pain, extremities (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT02489357/Prot_SAP_000.pdf